CLINICAL TRIAL: NCT07204418
Title: A Phase 1, 4-part, Open-label Study to Evaluate the Effects of CYP2D6 Phenotypes on the Pharmacokinetics of Xanomeline Following KarXT Administration in Healthy Adult Participants
Brief Title: A Study to Evaluate the Effects of CYP2D6 Phenotypes on the Pharmacokinetics of Xanomeline Following KarXT Administration in Healthy Adult Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Karuna Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CN012-0012
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteers
Keywords: Healthy volunteer; Pharmacokinetics; BMS-986510; KarXT; Cobenfy; CYP2D6
MeSH Terms: interventions — xanomeline; trospium chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- KarXT (Experimental)
  Interventions: Drug: Xanomeline/ Trospium Chloride

INTERVENTIONS:
Drug: Xanomeline/ Trospium Chloride — Specified dose on specified days
  Other Names: BMS-986510; KarXT

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (PK) of xanomeline following administration of KarXT in CYP2D6 normal/extensive, intermediate, poor, and ultrarapid metabolizers.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be healthy male and female (INOCBP) participants as determined by no clinically significant deviation from normal in medical history, physical examination, 12-lead electrocardiogram (ECG), vital signs (VS), and clinical laboratory determinations.
* Participant must be a normal/extensive, intermediate, poor, or ultrarapid CYP2D6 metabolizer.
* Participant must have body mass index (BMI) of 18.0 to 32.0 kg/m2, inclusive.

Exclusion Criteria:

* Participants must not have evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, 12-lead ECG, or clinical laboratory determinations beyond what is consistent with the target population reference ranges.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2026-12-03 (Estimated); Study Completion 2026-12-03 (Estimated)

PRIMARY OUTCOMES:
Geometric mean ratio for the area under the concentration-time curve from time zero to 12 hours post morning dose (AUC(0-12)) | Up to Day 17

SECONDARY OUTCOMES:
Number of participants with Adverse Events (AEs) | Up to 28 days post last dose
Number of participants with Serious Adverse Events (SAEs) | Up to 28 days post last dose
Number of participants with physical examination abnormalities | Up to 28 days post last dose
Number of participants with vital sign abnormalities | Up to 28 days post last dose
Number of participants with electrocardiogram (ECG) abnormalities | Up to 28 days post last dose
Number of participants with clinical laboratory test abnormalities | Up to 28 days post last dose
Columbia-Suicide Severity Rating Scale (C-SSRS) | Up to 28 days post last dose
Number of participants with AEs of Special Interest (AESIs) | Up to 28 days post last dose

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- United States (3):
  - Anaheim Clinical Trials, Anaheim, California
  - ICON - Lenexa, Lenexa, Kansas
  - ICON Development Solutions, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT07204418.html